CLINICAL TRIAL: NCT02534246
Title: A Paired Prospective, Single Blinded Study of the Diagnostic Accuracy and Specimen Adequacy of Two Endoscopic Tissue Biopsy Needles for Diagnosis Solid Pancreatic Mass
Brief Title: Head to Head Comparison of Two Needles EUS Guided FNB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, John M. Levenick, Assistance Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY2970
Record Dates: First submitted 2015-08-13; First posted 2015-08-27 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Pancreatic Tumor
Keywords: Core tissue biopsy; Core needle biopsy; EUS; Fine needle biopsy; Fine needle aspiration
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pro Core EUS guided Fine Needle Biopsy (Experimental): Echo Tip ProCore ultrasound biopsy needle (Cook Medical 25 gauge) with reverse bevel design for diagnosis of pancreatic lesions.
  Interventions: Device: Ultrasound biopsy needle Echo Tip ProCore
- Shark Core EUS guided Fine Needle Biopsy (Experimental): SharkCore ultrasound biopsy needle (Medtronic [Beacon] 25 gauge) with six cutting edge surfaces and an opposing bevel design for diagnosis of pancreatic lesions.
  Interventions: Device: Ultrasound biopsy needle SharkCore

INTERVENTIONS:
Device: Ultrasound biopsy needle Echo Tip ProCore — Two passes preformed with Echo Tip ProCore ultrasound biopsy needle (Cook Medical 25 gauge) and two passes will be performed using SharkCore ultrasound biopsy needle (Medtronic [Beacon] 25 gauge) from single lesion.
  Arms: Pro Core EUS guided Fine Needle Biopsy
Device: Ultrasound biopsy needle SharkCore
  Arms: Shark Core EUS guided Fine Needle Biopsy

SUMMARY:
The aim of this study is to evaluate and compare the diagnostic accuracy and specimen adequacy of two ultrasound biopsy needles. These are two existing FDA approved tissue biopsy regimens, with respect to diagnosis of solid pancreatic lesions.

DETAILED DESCRIPTION:
EUS guided core biopsy using various needle designs and sizes, seems to be a promising technique to procure tissue in solid pancreatic masses for making an accurate histological diagnosis. EUS-guided core biopsies of pancreas may aid in patients with non-diagnostic EUS-FNA samples and institutions where they do not have on-site cytopathology available for prompt evaluation of tissue adequacy. Making an accurate diagnosis not only assists in planning appropriate treatment but also may decrease morbidity/mortality from unnecessary surgeries.

Our goal is to evaluate and compare the diagnostic accuracy and specimen adequacy of the Cook Medical 25 gauge ProCore ultrasound biopsy needle and the Medtronic (Beacon) 25 gauge SharkCore ultrasound biopsy needle. We hypothesize the endoscopic ultrasound tissue biopsy will not be different in diagnostic accuracy of solid pancreatic lesions when using a 25 gauge SharkCore ultrasound biopsy needle in comparison with the 25 gauge ProCore ultrasound biopsy needle.

This is a non- inferior paired, prospective, single-blind study design in which patients undergoing EUS for a solid pancreatic mass. Two biopsies with each of the two endoscopic needles of interest in this study will be used in random order. The biopsy needle passed first will be randomized, after which the two needles will be alternated for each of the remaining biopsies. Randomization will occur in permuted blocks of 3. Physician will record the ease/ difficulty of obtaining each of the 4 biopsies on a scale of 1 to 5. Also, they record the needle visibility on ultrasound. The biopsy site will be examined for evidence of bleeding. Biopsies will be sent to the pathology laboratory in a blinded fashion in coded containers, where pathologist determine the number of adequate biopsies out of two passes of each needle.The pathologist will also provide a scale of perceived diagnostic usefulness of material in a blinded fashion. Post procedure care will including a letter to referring physician with recommendations for treatment and follow up.

This study include 30 patients referred to Hershey Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 18-90 of any gender, ethnicity and race that are referred to endoscopy for endoscopic ultrasound guided tissue acquisition for solid pancreatic mass.
* Voluntary enrollment
* Ability to give written informed consent
* Subjects must have a pancreatic mass detected by radiology (CT or MRI) or ultrasound or at the time of EUS.

Exclusion Criteria:

* Patients with coagulopathy with an elevated INR>2
* Any individual who cannot provide one's voluntary informed written consent.
* Any pre-existing or discovered medical condition that may at the discretion of investigator interfere with the completion of and/ or participation in existing protocol.
* Pregnancy
* Less than 18 years old

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Direct Comparison of pancreatic mass histologic tissue adequacy using two EUS guided fine needle biopsy needles | 1year
  Head to head comparison of tissue adequacy for solid pancreatic lesions using two 25 gauge EUS guided fine needle biopsy platforms - ProCore vs SharkCore.

CONTACTS AND LOCATIONS:
Overall Officials: John M Levenick, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States